CLINICAL TRIAL: NCT02818673
Title: Refractory Ascitis Diagnosis by the Study of Labelled Albumin Pharmacokinetics Between Peritoneal and Vascular Compartments
Brief Title: Refractory Ascitis Diagnosis by the Study of Labelled Albumin Pharmacokinetics
Acronym: ARAM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P140902; 2015-000157-20 (EudraCT Number)
Record Dates: First submitted 2016-06-20; First posted 2016-06-30 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Refractory Ascites in Patients With Cirrhosis
Keywords: diagnostic performances; ascites
MeSH Terms: conditions — Ascites | interventions — Iodine-125

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ascites in Patients With Cirrhosis (Experimental): Patients will be further classified according to the refractory or sensitive ascitis
  Interventions: Radiation: labelled human serumalbumin (125-I, Séralb®CisBio); Radiation: labelled albumin (99m-Tc, Vasculocis®, Cisbio)

INTERVENTIONS:
Radiation: labelled human serumalbumin (125-I, Séralb®CisBio) — Intra-veinous injection of 0,015 MBq/Kg ; 0,5 to 2 mL injected over less than a minute
Radiation: labelled albumin (99m-Tc, Vasculocis®, Cisbio) — intra-peritoneal injection of 200 MBq of labelled albumin (99m-Tc, Vasculocis®, Cisbio) ; 5 ml injected over less than a minute

SUMMARY:
Refractory ascites is an indication for liver transplantation, and includes ascites that is resistant to, or intractable by diuretic therapy (International Ascites Club). This definition is partly subjective; it can be established only a posteriori, following diuretic therapy administration to all patients, including those in whom untoward effects are prominent; and requires prolonged follow-up. An early diagnosis of refractory ascites would avoid giving diuretic therapy to patients in whom it will fail and identify rapidly candidates to liver transplantation. Such diagnosis could be done with a pharmacokinetic (PK) study of radiolabeled albumin between the peritoneal cavity and serum.

DETAILED DESCRIPTION:
Main objective: assess the performances of PK parameters (transfer of labelled albumin) between peritoneal and vascular compartments, for the diagnosis of refractory ascitis, in patients with cirrhosis and abundant ascitis.

Design: proof of concept study. Interventional cross-sectional study in Beaujon Hospital (Clichy, France), 1 recruiting center and 1 non recruiting center.

Patients are recruited in the Hepatology department (Pr Valla) and PK exploration is performed in the nuclear medicine department (Pr Lebtahi) of Beaujon Hospital.

Description of intervention: diuretics treatment discontinuation 7 days before exploration for patients with sensitive ascitis, and more than 7 days for those with refractory ascitis. The day of exploration, the patients come to hospital and stay in lying position. One intra-veinous injection of 0,015 megabecquerel(MBq) /Kg labelled human serum albumin (Iode-125 (125-I), Séralb®CisBio), in compliance with market authorization, simultaneously to one intra-peritoneal injection of 200 MBq of labelled albumin (Technetium 99m (99m-Tc), Vasculocis®, Cisbio), off-label used. It follows 5 minutes mobilization of the patient (right and left lateral decubitus), then a scintigraphy will be performed using a gamma-camera Symbia T2 (Siemens®). Repeated blood (5 ml) and peritoneal ascitis (3 ml) samples are performed before injection and every 30 minutes for 6 hours (catheter in place). Diuretic treatment can be restarted the day after PK explorations. Patients are followed-up at 1 month by phone call (for the collection of adverse events).

Measurements : radioactivity measurements of 99m-Tc and 125-I in the biological samples are performed by a counter device in the nuclear medicine department (Wizard 3000, Packard®). Unidirectional transfer of labelled albumin (125-I) from vascular compartment (plasma-P) to peritoneal compartment (ascitis-A) (TPA), Unidirectional transfer of labelled albumin (99m-Tc) from peritoneal (A) to vascular compartment (P) (TAP), and the ratio TPA/TAP are calculated from these measurements using Matlab®.The gold standard is defined by the diagnosis of refractory ascitis performed before inclusion.

Statistical analyses: performances of the TAP, of the TPA, and of the ratio TPA/TAP for the diagnosis of refractory ascitis, will be computed using the Receiver Operating Characteristic (ROC) curve.

Number of patients : 30 patients (15 patients with refractory ascitis and 15 patients with sensitive or untreatable ascitis) will be included during a 24 months period (1 or 2 patients per month), and followed-up for 2 months. The PK explorations will be performed in nuclear medicine department not more than 4 weeks after inclusion. Total length of study will be of 26 months.

ELIGIBILITY:
Inclusion Criteria:

* patients consulting in Hepatology department of Beaujon Hospital
* aged 18 - 80 years old
* cirrhosis due to alcoholic and/or dysmetabolic and/or viral (HBV or HCV) cause, pathologically or clinically/biologically/radiologically proven.
* Volume of ascitis >5 L, either sensible or refractory to diuretics drugs according IAC criteria

Exclusion Criteria:

* infection in the 2 weeks prior to inclusion (suspected or proven)
* upper gastrointestinal bleeding du to portal hypertension in the 2 weeks prior to inclusion
* transjugular intrahepatic portosystemic shunt (TIPS)
* advanced hepatocellular carcinoma
* hepatic transplantation
* unability to stay lying for 6 hours
* pregnancy / lactation
* renal deficiency (creat. clearance < 60ml/min)
* cardiac deficiency (≥ New York Heart Association (NYHA) III) or myocardial infarction (<3 months)
* other cause of ascitis
* contra-indication to human albumin (125-I) or vasculosis (99m-Tc) or other component of radio-pharmaceutics
* no health insurance coverage
* unability to go to the hospital for 1 day of exams
* refuse to consent to study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of refractory ascitis according to International Ascites Club (IAC) | Exploration day (4 weeks after the inclusion)

SECONDARY OUTCOMES:
Measure of pharmacokinetics parameters : TPA | Exploration day (4 weeks after the inclusion)
  radioactivity measurements of labelled albumin (125-I) in ascitis (peritoneal samples) and plasma (blood samples)
Measure of pharmacokinetics parameters : TAP | Exploration day (4 weeks after the inclusion)
  radioactivity measurements of labelled albumin (99m-Tc) in ascitis (peritoneal samples) and plasma (blood samples)
Measure of pharmacokinetics parameters | Exploration day (4 weeks after the inclusion)
  Ratio TPA/TAP
adverse events | 1 month after exploration day
  Phone call
Proportion of patients in whom examination conditions and technical feasibility were completed | Exploration day (4 weeks after the inclusion)
  adequate volume of ascites,stable state of patient, satisfactory spread of radiopharmaceuticals in the peritoneal compartment measure by scintigraphy, number of peritoneal and blood samples performed

CONTACTS AND LOCATIONS:
Overall Officials: VALLA Dominique, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Beaujon, Clichy, France

IPD SHARING:
Plan to Share IPD: Undecided